CLINICAL TRIAL: NCT05823519
Title: Neck Evolution With Ovation in Spain
Acronym: NEOVAS
Status: Recruiting | Type: Observational
Sponsor: DGM Vascular (Network)
Collaborators: Hospital Universitario Central de Asturias (Other)
Responsible Party: Sponsor
Other Study IDs: NEOVAS
Record Dates: First submitted 2023-03-14; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Alto Endograft; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- SINGLE Arm: Observational, Multicenter, Prospective, single arm registry study with consecutive, eligible patient enrollment at each site. Subjects will be followed procedurally to discharge, and as per institutional standard of care thereafter through to 3 years (total follow-up commitment), with follow up including Computed tomography angiography (CTA) study and Case Report Form data at 1 month, 6 months, 1 years, 2 years and 3 years, closing at this time the study primary endpoint.
  Interventions: Device: Endologix Ovation Alto Endograft

INTERVENTIONS:
Device: Endologix Ovation Alto Endograft — Implantation of aorto-bisiliac ALTO endograft to exclude Abdominal Aortic Aneurysms

SUMMARY:
This is a multicenter, observational, prospective, single arm registry using Ovation Alto Endograft. A minimum of 50 up to a maximum of 120 subjects undergoing endovascular repair with Ovation Alto endograft will be enrolled and followed procedurally to discharge, at 1month, 6 months, 1 year and yearly afterward up to 3 years. This registry of Ovation Alto endograft will provide further assessment to confirm continuing safety and effectiveness of the graft and to confirm the stability of the neck diameter over time when treated with this device.

DETAILED DESCRIPTION:
Abdominal Aortic Aneurysm (AAA) is a widespread disease with a high mortality rate in case of ruptures, with a sizable number of patients dying before a diagnosis is made. Approximately 32.000 patients are newly diagnosed with AAA and about 44.000 repair procedures are performed in the US every year. It is estimated that up to 2.000.000 subjects are living with an undiagnosed AAA with a greater incidence in the elderly population >65 years. Risk factors include smoking, hypertension, hypercholesterolemia, gender (men/women ratio 5:1) and family history (15-20%) increase risk amongst first degree relatives. The rupture risk increases with age and concomitant hypertension as well as current tobacco use and presence of other cardio-vascular diseases. AAA is clinically defined as a focal dilatation of the aorta causing a diameter increase of >50% of the expected normal diameter. Although any artery may develop an aneurysm, they are most commonly observed in the infrarenal abdominal aorta, thoracic aorta, popliteal artery and common iliac artery. The concomitants risks related to aneurysms are rupture and thrombus migration. Aneurysms slowly and continually grow in size leading to the aneurysm bursts. The larger an aneurysm becomes, the likelihood of eventual rupture may appear. The natural outcomes of aortic aneurysms is to enlarge and rupture. Other potential complications of the aneurysm include compression of adjacent organs which may result in aortoenteric fistula, or aortocaval fistula. If the thrombus embolizes and flows down the blood stream, this can induce acute or chronic arterial obliteration of the lower limbs.The risk of rupture is weighed against the risk of perioperative morbidity. The United Kingdom Small Aneurysm trial (UKSAT) reported 103 aneurysm ruptures in 2,257 subjects over a period of seven years, with an annual rupture rate of 2.2%. The decision to treat a patient that presents with an asymptomatic aneurysm is primarily dependent upon the size of the aneurysm. Current Society for Vascular Surgery (SVS) practice guidelines recommend surveillance for most subjects with a fusiform AAA in the range of 4.0 to 5.4cm in maximum diameter; therefore, surgical repair of abdominal aneurysms of 5.5 cm or greater in diameter is recommended in healthy subjects, as it is repair of saccular aneurysms. With the development of endovascular treatment options in recent years, treatment of AAA has become a viable option for patients with a high pre-operative risk. Endovascular Aneurysm Repair (EVAR) has become the treatment strategy of choice for AAA. Nowadays, the most important limit to the effectiveness of this technique is represented by complex anatomical situations, especially regarding the morphology of the proximal sealing zone. In previously published studies, the use of EVAR outside the specific instructions for use (IFU) of the devices for patients with challenging proximal aortic necks yielded a non-negligible rate of immediate complications and re-interventions. The Ovation iX and Alto endografts represent a new technical step in EVAR. This new device separates fixation from sealing: fixation is guaranteed by suprarenal stent and anchors, while sealing is ensured by inflatable rings filled with a low-viscosity, non-embolic, radiopaque fill polymer. This unique characteristic allows this graft to isolate aortic neck from blood pressure without radial force, with the result of very low ratios of Type 1 Endoleaks and absence aortic neck growing. The presence of the polymer-filled network also allows the graft to conform to the patient's aortic neck, providing precise and reliable sealing in a great variety of anatomies. Different from common stent-graft platforms, separation between fixation and sealing ensures that stent and fabric do not compete in the Ovation endograft for the same space within the shaft, and an ultra-low-profile delivery system can be achieved, allowing the treatment of patients presenting a wide range of iliac access.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years old.
2. Subject has signed informed consent for data release.
3. Subjects with de novo infrarenal AAA /aorto-iliac AAA and eligible for endovascular Abdominal Aortic Aneurysm Repair with the Ovation Alto Endograft according to current IFU.

Exclusion Criteria:

1. Currently participating in another study where primary endpoint has not been reached yet.
2. Currently participating in another study with the same devices and/or the same primary endpoint.
3. Known allergy to any of the device components.
4. Pregnant (females of childbearing potential only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female at least 18 years old with aortic abdominal aneurysm with characteristics within the IFU of de device
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Post-implant infrarenal aneurysm's neck grow evaluation | 30 days
  The neck diameter will be measured on Computed Tomography Angiography (CTA) at 0mm (lowest renal artery), 5mm, 10mm, 15mm and 20mm. No type I or III endoleak. No clinically significant migration (>5mm). No Aneurysm enlargement (>5mm)
Post-implant infrarenal aneurysm's neck grow evaluation | 6 months
  The neck diameter will be measured on Computed Tomography Angiography (CTA) at 0mm (lowest renal artery), 5mm, 10mm, 15mm and 20mm. No type I or III endoleak. No clinically significant migration (>5mm). No Aneurysm enlargement (>5mm)
Post-implant infrarenal aneurysm's neck grow evaluation | 1 year
  The neck diameter will be measured on Computed Tomography Angiography (CTA) at 0mm (lowest renal artery), 5mm, 10mm, 15mm and 20mm. No type I or III endoleak. No clinically significant migration (>5mm). No Aneurysm enlargement (>5mm)
Post-implant infrarenal aneurysm's neck grow evaluation | 2 years
  The neck diameter will be measured on Computed Tomography Angiography (CTA) at 0mm (lowest renal artery), 5mm, 10mm, 15mm and 20mm. No type I or III endoleak. No clinically significant migration (>5mm). No Aneurysm enlargement (>5mm)
Post-implant infrarenal aneurysm's neck grow evaluation | 3 years
  The neck diameter will be measured on Computed Tomography Angiography (CTA) at 0mm (lowest renal artery), 5mm, 10mm, 15mm and 20mm. No type I or III endoleak. No clinically significant migration (>5mm). No Aneurysm enlargement (>5mm)

SECONDARY OUTCOMES:
Procedural technical success | Immediately after the procedure
  Immediate procedural technical success
Aneurysm evaluation | 3 years
  No Aneurysm rupture
Related mortality | 3 years
  AAA-related mortality
Secondary Evaluations | 3 years
  Conversion to open surgical
Polymer leak | 3 years
  No polymer leak during and after implant

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Alonso Pérez, MD, Principal Investigator — Hospital Universitario Central de Asturias
Locations (9):
- Spain (9):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario De Girona Dr. Josep Trueta, Girona, Barcelona
  - Hospital Universitario De Cruces, Barakaldo, Bizkaia
  - Hospital Universitario De Burgos, Burgos, Castille and León
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital General Universitario De Toledo, Toledo, Castille-La Mancha
  - Hospital Universitario De Cabueñes, Gijón, Principality of Asturias
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona

IPD SHARING:
Plan to Share IPD: No